CLINICAL TRIAL: NCT02684812
Title: Ultra-early Tranexamic Acid After Subarachnoid Hemorrhage. A Prospective, Randomized, Multicenter Study.
Brief Title: Ultra-early Tranexamic Acid After Subarachnoid Hemorrhage.
Acronym: ULTRA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Stichting Nuts Ohra (Other)
Responsible Party: Principal Investigator, R. Post, Drs., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-000343-26
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Subarachnoid Hemorrhage
Keywords: antifibrinolytic therapy; recurrent bleeding; tranexamic acid
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: PROBE Design
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Active Comparator): Eligible subjects are randomly assigned to immediate administration of TXA (1 g i.v.) after a diagnosis of SAH, as confirmed by CT-scan of the brain, continued by continuous infusion of 1 g per 8 hours to a maximum of 24 hours after start of medication. A maximum of 4 g TXA (1 g bolus + 3x 1 g continuous infusion) can be administered to one patient.
  Interventions: Drug: Tranexamic Acid
- Control (No Intervention): Standard care

INTERVENTIONS:
Drug: Tranexamic Acid — Treatment until aneurysm treatment or maximum dosage of 4 gram
  Other Names: Cyklokapron
  Arms: Tranexamic Acid

SUMMARY:
This is a multicenter, prospective, randomized, open-label trial with blinded endpoint (PROBE) assessment. Adult patients with the diagnosis of non-traumatic SAH, as proven by computed tomography (CT) within 24 hours after the onset of headache, will be randomly assigned to the treatment group or the control group. Patients in the treatment group will receive standard treatment with the addition of a bolus of TXA (1 g intravenously) immediately after randomization, followed by continuous infusion of 1 g per 8 hours until the start of aneurysm treatment, or a maximum of 24 hours after the start of medication. Patients in the control group will receive standard treatment without TXA. The primary outcome measure is favorable functional outcome, defined as a score of 0 to 3 on the modified Rankin Scale (mRS), at 6 months after SAH. Primary outcome will be determined by a trial nurse blinded for treatment allocation.

DETAILED DESCRIPTION:
Approximately 50% of all patients with a subarachnoid hemorrhage (SAH) die due to the hemorrhage or subsequent complications. There are several major causes for this course, such as in-hospital rebleed in 21.5% which most frequently occurs within the first 6 hours after the primary hemorrhage ("ultra-early rebleed"). A major part of the patients with a rebleed die during hospital admission and when they survive, they develop more severe cognitive dysfunctions. Reducing the rebleeds by ultra-early administration of tranexamic acid (TXA) could be a major factor in improving the functional outcome after SAH.

To evaluate whether SAH patients treated by state-of-the-art SAH management with additional ultra-early and short term TXA administration have a significantly higher percentage of favourable outcome after six months (score 0-3 on the Modified Rankin Scale) compared to the group treated by up-to-date SAH management without additional TXA.

To evaluate whether: 1) TXA reduces in-hospital rebleeds and case fatalities; 2) TXA causes more ischemic stroke 3) TXA causes more complications (such as thromboembolic events, hydrocephalus, extracranial thrombosis or hemorrhagic complications) during treatment, admission and follow-up; 4) there is a difference in causes of poor outcome between groups; 5) there is a difference in discharge locations between groups; 6) there is an association between the time between hemorrhage and TXA administration and outcome; 7) TXA increases (micro)infarctions after endovascular treatment; 8) TXA reduces health-care costs between discharge and six months after hemorrhage; 9) TXA improves quality of life at six months after hemorrhage; 10) there are differences in rebleed rates and outcome between genders or groups with different WFNS scores at admission.

Multicenter, prospective, randomized, open label treatment with blind endpoint assessment.

Adult patients (18 years and older) included within 24 hours after SAH. Group one: standard treatment with additional administration of 1 g TXA intravenously in ten minutes, immediately after the diagnosis SAH, succeeded by continuous infusion of 1 g per 8 hours until a maximum of 24 hours. Group two: standard treatment with no TXA administration. Both groups undergo a standardized and validated interview at discharge and six months after hemorrhage to assess the modified Rankin Scale score, and both groups receive a questionnaire to evaluate health-care costs and quality of life.

Primary: modified Rankin Scale score after six months, dichotomized into favourable and unfavourable outcome. Secondary: rebleed and case fatality rate, complications during the first six months after hemorrhage, (micro)infarctions at MR imaging after endovascular treatment, health-care costs from discharge until six months, quality of life at six months and differences in rebleed rates and outcome between genders or WFNS score at admission.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects are randomly allocated to ultra-early TXA therapy or standard treatment. Complications are minor and the expected benefit is large compared with separate studies done with antifibrinolytic medications. In these studies, the safety of the use of these medications in this study population is confirmed. In this patient group there are adequate, disoriented and comatose patients on admission, so a part of the studied patients are incapacitated when undergoing the study. To extrapolate the conclusions of this study to clinical protocols it is necessary to include patients with a SAH in all different severity grades. Weighing carefully the benefits versus the burden and risks, it is assumed that patients will benefit from ultra-early TXA administration with minimal burden during therapy.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the study centers or their referring hospitals
* CT-confirmed SAH with most recent ictus less than 24 hours ago Definition: subarachnoid hemorrhage is a bleeding pattern on computed tomography with hyperdensity in the basal cisterns and/or Sylvian or interhemipheric fissures or a intraparenchymal hyperdensity consistent with a hematoma from an anterior, a pericallosal, a posterior or a middle cerebral artery aneurysm.

Exclusion Criteria:

* No proficiency of the Dutch or English language
* No loss of consciousness after the hemorrhage with WFNS grade 1 or 2 on admission in combination with a perimesencephalic hemorrhage Definition: on CT examination presence of hyperdensities exclusively in the basal cisterns maximal extending to the proximal part of the Sylvian fissure or posterior part of the interhemispheric fissure, without evidence for intracerebral or intraventricular haemorrhage (except slight sedimentation)
* Bleeding pattern on CT compatible with a traumatic SAH
* Treatment for deep vein thrombosis or pulmonary embolism
* History of a blood coagulation disorder (a hypercoagulability disorder)
* Pregnancy checked with a pregnancy test in women in their childbearing period
* History of severe renal (serum creatinin >150 mmol/L)
* History of severe liver failure (AST > 150 U/l or ALT > 150 U/l or AF > 150 U/l or γ-GT > 150 U/l)
* Imminent death within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | six months
  Good (mRS 0-3) and Poor (mRS 4-6)

SECONDARY OUTCOMES:
Date and cause of death | Maximum six month
  Assessment of cause of death by a committee (intensive care/neurosurgeon)
Cause of poor outcome | six months
  Assessment of which events during hospital admission led to a poor outcome defined as mRS 4 and 5 by a committee (intensive care/neurosurgeon)
Rebleed and time interval after first hemorrhage | six months
  The time interval between the initial hemorrhage and occurence of a recurrent bleeding will be recorded.
Thromboembolic events during endovascular treatment | up to 48 hours
  Complications during endovascular treatment will be recorded (ie occurence of clotting in one of the vessels)
Ischemic stroke (Dealyed cerebral ischemia) | 14-20 days
Extracranial thrombosis | six months
Hydrocephalus and treatment modality | six months
  Occurence of a hydrocephalus will be recorded and which treatment modality is used to treat the hydrocephalus
Hemorrhagic complications (intra- and extracranial) | six months
Time interval from last hemorrhage to first TXA administration | 24 hours
Discharge location | six months
Infarctions on MR imaging at six months after endovascular treatment | six months
Health-care costs between discharge and six months after hemorrhage | three and six months
  Questionnaires
Quality of life at six months after hemorrhage | six months
  Questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: William P Vandertop, PhD MD, Principal Investigator — Department of Neurosurgery
Locations (1):
- Academic Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Germans MR, Post R, Coert BA, Rinkel GJ, Vandertop WP, Verbaan D. Ultra-early tranexamic acid after subarachnoid hemorrhage (ULTRA): study protocol for a randomized controlled trial. Trials. 2013 May 16;14:143. doi: 10.1186/1745-6215-14-143. PMID 23680226
- [Derived] Denneman N, Post R, van Eekelen R, Tjerkstra MA, Kempeneers MA, Labib H, Germans MR, Vergouwen MDI, Jellema K, Koot RW, Kruyt ND, Wolfs JFC, Nanda D, Van Der Pol B, Roks G, De Beer F, Reichman LJA, Brouwers PJAM, Vincent HK 1st, Bienfait HP, Boogaarts HD, Klijn CJM, van den Berg R, Coert BA, Horn J, Majoie CBLM, Rinkel GJE, Roos YBWEM, Vandertop WP, Verbaan D; ULTRA trial study group. Cost-Effectiveness of Ultra-Early Tranexamic Acid as Add-On to Standard Care After Subarachnoid Hemorrhage (ULTRA Trial). Eur J Neurol. 2025 Aug;32(8):e70208. doi: 10.1111/ene.70208. PMID 40843772
- [Derived] Tjerkstra MA, Post R, Germans MR, Vergouwen MDI, Jellema K, Koot RW, Kruyt ND, Wolfs JFC, De Beer FC, Kieft HH, Nanda D, Van Der Pol B, Roks G, De Beer F, Reichman LJA, Brouwers PJAM, Kwa VIH, Van Der Ree TC, Bienfait HP, Boogaarts HD, Klijn CJ, Visser V, van den Berg R, Coert BA, Horn J, Majoie CBLM, Rinkel GJE, Roos YBWEM, Vandertop WP, Verbaan D; ULTRA trial study group. Ultra-Early and Short-Term Tranexamic Acid Treatment in Patients With Good- and Poor-Grade Aneurysmal Subarachnoid Hemorrhage. Neurology. 2024 Jun 25;102(12):e209169. doi: 10.1212/WNL.0000000000209169. Epub 2024 May 24. PMID 38788175
- [Derived] Vergouwen MD, Germans MR, Post R, Tjerkstra MA, Coert BA, Rinkel GJ, Peter Vandertop W, Verbaan D. Aneurysm treatment within 6 h versus 6-24 h after rupture in patients with subarachnoid hemorrhage. Eur Stroke J. 2023 Sep;8(3):802-807. doi: 10.1177/23969873231173273. Epub 2023 May 1. PMID 37641555
- [Derived] Tjerkstra MA, Post R, Germans MR, Vergouwen MDI, Jellema K, Koot RW, Kruyt ND, Willems PWA, Wolfs JFC, de Beer FC, Kieft H, Nanda D, van der Pol B, Roks G, de Beer F, Halkes PHA, Reichman LJA, Brouwers PJAM, Van den Berg-Vos RM, Kwa VIH, van der Ree TC, Bronner I, Bienfait HP, Boogaarts H, Klijn CJM, van den Berg R, Coert BA, Horn J, Majoie CBLM, Rinkel GJE, Roos YBWM, Vandertop WP, Verbaan D; ULTRA investigators. Tranexamic Acid After Aneurysmal Subarachnoid Hemorrhage: Post Hoc Analysis of the ULTRA Trial. Neurology. 2022 Dec 5;99(23):e2605-e2614. doi: 10.1212/WNL.0000000000201160. PMID 36266046
- [Derived] Post R, Germans MR, Tjerkstra MA, Vergouwen MDI, Jellema K, Koot RW, Kruyt ND, Willems PWA, Wolfs JFC, de Beer FC, Kieft H, Nanda D, van der Pol B, Roks G, de Beer F, Halkes PHA, Reichman LJA, Brouwers PJAM, van den Berg-Vos RM, Kwa VIH, van der Ree TC, Bronner I, van de Vlekkert J, Bienfait HP, Boogaarts HD, Klijn CJM, van den Berg R, Coert BA, Horn J, Majoie CBLM, Rinkel GJE, Roos YBWEM, Vandertop WP, Verbaan D; ULTRA Investigators. Ultra-early tranexamic acid after subarachnoid haemorrhage (ULTRA): a randomised controlled trial. Lancet. 2021 Jan 9;397(10269):112-118. doi: 10.1016/S0140-6736(20)32518-6. Epub 2020 Dec 23. PMID 33357465
- [Derived] Post R, Germans MR, Coert BA, Rinkel GJE, Vandertop WP, Verbaan D. Update of the ULtra-early TRranexamic Acid after Subarachnoid Hemorrhage (ULTRA) trial: statistical analysis plan. Trials. 2020 Feb 18;21(1):199. doi: 10.1186/s13063-020-4118-5. PMID 32070395